CLINICAL TRIAL: NCT04832646
Title: VOLTage Mapping in Atrial Fibrillation
Acronym: VOLT-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GUENANCIA Charles, Associate Professor, Central Hospital, Nancy, France
Other Study IDs: 2020PI262
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation, Persistent
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: atrial fibrillation ablation — persistent atrial fibrillation ablation with both AF and sinus rhythm map available

SUMMARY:
The purpose of this study is to retrospectively analyze electroanatomical data collected during persistent atrial fibrillation ablation procedures, combined with pre-ablation cardiac CT data, in order to:

* define a new method for quantifying left atrial voltage in atrial fibrillation via a total energy map instead of a peak-to-peak amplitude map
* confirm the association between epicardial fat localization and atrial conduction slowing

DETAILED DESCRIPTION:
Background:

Atrial fibrillation (AF) is the most common arrhythmia, with an estimated prevalence in 2010 of 33.5 million people (3% of the world population). It is now estimated that 1 in 4 middle-aged adults in Europe and the United States will develop AF in their lifetime. Of course, the aging of the population is considered one of the major explanations for this pandemic phenomenon, as well as the ever-increasing prevalence of overweight and obesity. Complications related to this arrhythmia are numerous and frequent, with thromboembolic events having a major impact on morbidity. Thus, it is estimated that AF is responsible for a quarter of ischemic strokes and increases the risk of stroke fivefold. At the same time, there is an increased risk of long-term heart failure, which is responsible for excess mortality. Finally, patients with AF frequently have an impaired quality of life and a higher rate of hospitalization than patients in sinus rhythm (10 to 40% of patients with AF are hospitalized at least once a year). An association between AF and cognitive decline and risk of vascular dementia (even in patients treated with anticoagulants) has also been described. Depending on the temporality of AF, it is referred to as paroxysmal, persistent, or permanent AF.

Endocavitary ablation for the treatment of atrial fibrillation was first described by the Bordeaux team of Prof. Michel Haïssaguerre in the early 1990s, who demonstrated the role of electrical discharges from the pulmonary veins in the initiation of (paroxysmal) AF. The following years therefore saw the development of tools to electrically isolate the pulmonary veins from the left atrium, and then to try to identify and treat additional pathological areas in the atria for more advanced (persistent) forms of AF. The advent of three-dimensional modeling technologies has made it possible to develop intracardiac navigation systems to guide AF ablation in 3D, while limiting fluoroscopy time for the patient and staff.

In persistent AF, unlike paroxysmal AF, the technique used and the ablation targets are less codified, with success rates lower than those obtained in paroxysmal AF. Indeed, unlike paroxysmal AF, the pathophysiology of which is well understood, there is no unicist consensus theory for persistent AF. Based on the hypothesis of the predominance of the substrate over the pulmonary venous trigger in the self-maintenance of persistent AF, teams have highlighted the major role of left atrial fibrosis in this pathology, which is the cause of conduction heterogeneity in the left atrium. Work to elucidate the triggers of this fibrotic disease emphasizes the key role of periatrial epicardial fat, which secretes pro-fibrotic mediators and deregulates the atrial ganglionic plexi. An association has also been made between epicardial fat volume and the incidence and maintenance of atrial fibrillation. In addition, recent work demonstrates that the peri-atrial adipocyte environment modulates not only fibrosis but also the conductive properties of atrial cells.

During endocavitary ablation of atrial fibrillation, multi-electrode diagnostic catheters allow precise electroanatomical reconstruction of the left atrium, quantifying its geometry but also the local electrical signals (electrograms), in terms of amplitude (voltage map) and temporality relative to a reference (activation map). It is therefore theoretically possible to build a map of conduction velocities in sinus rhythm or electroentrainment in the atrium, by calculating the velocity and vector of electrical depolarization between each electrogram. In parallel, before any AF ablation, an injected cardiac CT scan is performed for three-dimensional atrial reconstruction. This scan also allows the quantification of the atrial epicardial fat in terms of volume and density. We therefore want to develop an algorithm allowing the construction of a map of velocities in sinus rhythm, fused to the three-dimensional reconstruction of the location of the atrial epicardial fat.

ELIGIBILITY:
Inclusion Criteria:

* Persistant Atrial fibrillation ablation
* Voltage map in sinus rhythm and in atrial fibrillation
* Cardiac CT scan performed before ablation

Exclusion Criteria:

* Incomplete data, poor quality ECG recordings.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted for a procedure in the interventional electrophysiology department of the CHRU de Nancy for AF ablation between March 2019 and March 2021, for whom electroanatomical and scannographic data are available
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
correlation between voltage map in sinus rhythm and the new voltage map in atrial fibrillation using total energy calculation | through study completion, an average of 1 year

SECONDARY OUTCOMES:
correlation between atrial epicardial fat deposits and atrial conduction velocities slowing | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Charles GUENANCIA, MD, PhD, Principal Investigator — CHRU Nancy
Locations (1):
- University Hospital of Nancy, Vandœuvre-lès-Nancy, France